CLINICAL TRIAL: NCT02906020
Title: Multicenter, Randomized, Double-blind, Placebo Controlled Study to Assess the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of GZ/SAR402671 in Patients With Early-stage Parkinson's Disease Carrying a GBA Mutation or Other Pre-specified Variant
Brief Title: A Global Study to Assess the Drug Dynamics, Efficacy, and Safety of Venglustat (GZ/SAR402671) in Parkinson's Disease Patients Carrying a Glucocerebrosidase (GBA) Gene Mutation
Acronym: MOVES-PD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The topline results of the 52-week double-blind placebo-controlled period were analyzed. The study did not meet the primary or secondary endpoints. Based on these results, the decision was made to halt the long-term follow-up period of the study
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT14820; 2016-000657-12 (EudraCT Number); U1111-1180-6918 (Registry Identifier: ICTRP)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2022-02-28 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — venglustat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GZ/SAR402671 (Experimental): Part 1: Increasing doses of GZ/SAR402671 were administered once per day. Part 2: A dose of GZ/SAR402671 (determined in Part 1) was administered once per day.
  Interventions: Drug: venglustat GZ/SAR402671
- Placebo (Placebo Comparator): A matching placebo for Parts 1 and 2 was administered once per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: venglustat GZ/SAR402671 — Pharmaceutical form: capsule Route of administration: oral
  Arms: GZ/SAR402671
Drug: Placebo — Pharmaceutical form: capsule Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objectives:

* Part 1: To determine the safety and tolerability of 4, 8, and 15 milligrams of GZ/SAR402671 (venglustat) administered orally for 4 weeks, as compared to placebo in participants with early-stage Parkinson's disease (PD) carrying a glucocerebrosidase gene (GBA) mutation or other pre-specified variants.
* Part 2: To determine the efficacy of GZ/SAR402671 administered orally daily, as compared to placebo in participants with early-stage PD carrying a GBA mutation or other pre-specified variants.

Secondary Objectives:

Part 1:

* To assess the pharmacokinetic (PK) profile of oral dosing of GZ/SAR402671 in plasma when administered in early-stage PD participants carrying a GBA mutation.
* To assess the exposure of GZ/SAR402671 in cerebrospinal fluid (CSF) when administered in early-stage PD participants carrying a GBA mutation.

Part 2:

* To demonstrate overall safety and tolerability of GZ/SAR402671 administered orally for 52 weeks in early-stage PD participants carrying a GBA mutation as compared to placebo.
* To assess the pharmacodynamic response to daily oral dosing of GZ/SAR402671 in plasma and CSF as measured by glucosylceramide (GL-1) when administered in early-stage PD participants carrying a GBA mutation over a 52-week period.

DETAILED DESCRIPTION:
Part 1: the total duration was as following:

i) Rest of the world (ROW): up to approximately 50 weeks (8.5 weeks of screening, maximum of 36 weeks of treatment and 6 weeks follow-up).

ii) Japan only: up to approximately 66 weeks (8.5 weeks of screening, maximum of 52 weeks of treatment and 6 weeks follow-up).

Part 2: the total duration was up to approximately 224 weeks that consisted of 8.5 weeks of screening period, 52 weeks of treatment period, 156 weeks of long-term follow-up (LTFU) period and 8 weeks of post-treatment period.

At the end of a 52-week main placebo-controlled treatment period, all participants were evaluated for possibility to transition to receive active treatment for 156 weeks plus 8-week post-treatment observation.

ELIGIBILITY:
Inclusion criteria:

* Male and female adults with a diagnosis of PD and who were heterozygous carriers of a GBA mutation associated with PD.
* Participants carrying known sequence variants associated with GBA-PD must had rapid eye movement (REM) sleep behavior disorder (RBD) confirmed by historically documented polysomnography or by questionnaire.
* Age greater than or equal to (>=) 18 years to 80 years inclusive at the time of informed consent signing (FOR JAPANESE PARTICIPANTS ONLY: Age >=20 years to 80 years, inclusive, at the time of signing the informed consent. Note: Japanese participants refers only to Japanese participants enrolled and living in Japan).
* Had symptoms of PD >=2 years.
* Hoehn and Yahr (H and Y) stage of 2 or lower at baseline.
* Stable medication regimen of PD drugs for at least 30 days (at least 60 days for rasagiline) prior to randomization.
* The participant was willing to abstain from grapefruit containing products for 72 hours prior to administration of the first dose of GZ/SAR402671 and for the duration of the entire treatment period (Part 1 and Part 2, Periods 2 and 3).
* Signed written consent.

Exclusion criteria:

* Parkinsonism due to drug(s) or toxin(s).
* Participants carrying the LRRK2 G2019S mutation.
* Participants with Gaucher disease (GD) as defined by clinical signs and symptoms (i.e., hepatosplenomegaly, cytopenia, skeletal disease) and/or marked deficiency of GCase activity compatible with GD.
* Montreal Cognitive Assessment score less than 20.
* Participants with prior surgical history of deep brain stimulation (DBS).
* Participants with baseline brain MRI without contrast showing a structural abnormality that is a possible cause of their PD signs or symptoms.
* Hepatic insufficiency with liver function tests (LFT) greater than (>) 2 times upper limit of normal at Screening Visit.
* The participant had a documented diagnosis, as per local regulations, of any of the following infections: hepatitis B, hepatitis C, human immunodeficiency virus 1 or 2.
* Renal insufficiency as defined by creatine >1.5 times normal at Screening Visit.
* The participant had received strong or moderate inducers or inhibitors of CYP3A4 within 30 days or 5 half-lives prior to randomization, whichever is longer.
* The participant had, according to World Health Organization (WHO) Grading, a cortical cataract > one-quarter the lens circumference (grade cortical catact-2 [COR-2]) or a posterior subcapsular cataract >2 millimeters (grade posterior subscapsular cataract [PSC-2]). Participant with nuclear cataracts would not be excluded.
* The participant was currently receiving potentially cataractogenic medications, including chronic regimen (more frequently than every 2 weeks) of any dose or route of corticosteroids or any medication that could cause cataract or worsen the vision of participants with cataract (eg, glaucoma medications) according to the Prescribing Information.
* If female, pregnant (defined as positive beta-human chorionic gonadotrophin [Beta-HCG] blood test) or lactating or breast-feeding.
* Any medical disorders and/or clinically relevant findings that, in the opinion of the Investigator, could interfere with study-related procedures. This included condition(s) that precluded the safe performance of routine lumbar punctures, such as prohibitive spinal diseases, bleeding diasthesis, or clinically significant coagulopathy or thrombocytopenia.
* Current participation in another investigational interventional study.
* Any medications specifically used for treating memory dysfunction, such as, but not limited to cholinesterase inhibitors or memantine, within 30 days or 5 half-lives of these medications prior to randomization, whichever was longer.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (52):
- United States (19):
  - Investigational Site Number :8400017, Scottsdale, Arizona
  - Investigational Site Number :8400011, Scottsdale, Arizona
  - Investigational Site Number :8400004, La Jolla, California
  - Investigational Site Number :8400019, Palo Alto, California
  - Investigational Site Number :8400013, Sunnyvale, California
  - Investigational Site Number :8400015, New Haven, Connecticut
  - Investigational Site Number :8400008, Boca Raton, Florida
  - Investigational Site Number :8400016, Chicago, Illinois
  - Investigational Site Number :8400005, Chicago, Illinois
  - Investigational Site Number :8400014, Boston, Massachusetts
  - Investigational Site Number :8400018, New York, New York
  - Investigational Site Number :8400010, New York, New York
  - Investigational Site Number :8400001, New York, New York
  - Investigational Site Number :8400021, Portland, Oregon
  - Investigational Site Number :8400020, Portland, Oregon
  - Investigational Site Number :8400009, Portland, Oregon
  - Investigational Site Number :8400002, Philadelphia, Pennsylvania
  - Investigational Site Number :8400006, Fairfax, Virginia
  - Investigational Site Number :8400012, Kirkland, Washington
- Investigational Site Number :0400001, Innsbruck, Austria
- Canada (3):
  - Investigational Site Number :1240003, Vancouver, British Columbia
  - Investigational Site Number :1240002, Ottawa, Ontario
  - Investigational Site Number :1240001, Montreal, Quebec
- Investigational Site Number :2500001, Paris, France
- Germany (2):
  - Investigational Site Number :2760002, Kiel
  - Investigational Site Number :2760001, Tübingen
- Investigational Site Number :3000002, Larissa, Greece
- Israel (4):
  - Investigational Site Number :3760002, Haifa
  - Investigational Site Number :3760003, Petah Tikva
  - Investigational Site Number :3760001, Tel Aviv
  - Investigational Site Number :3760004, Tel Litwinsky
- Italy (5):
  - Investigational Site Number :3800006, Rozzano, Milano
  - Investigational Site Number :3800001, Catanzaro
  - Investigational Site Number :3800004, Milan
  - Investigational Site Number :3800003, Pavia
  - Investigational Site Number :3800002, Salerno
- Japan (5):
  - Investigational Site Number :3920005, Nagoya, Aichi-ken
  - Investigational Site Number :3920002, Kyoto, Kyoto
  - Investigational Site Number :3920004, Osaka, Osaka
  - Investigational Site Number :3920001, Bunkyo-ku, Tokyo
  - Investigational Site Number :3920003, Kodaira-shi, Tokyo
- Investigational Site Number :5780001, Trondheim, Norway
- Portugal (2):
  - Investigational Site Number :6200002, Coimbra
  - Investigational Site Number :6200003, Torres Vedras
- Singapore (2):
  - Investigational Site Number :7020001, Singapore
  - Investigational Site Number :7020002, Singapore
- Spain (2):
  - Investigational Site Number :7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240001, Seville
- Investigational Site Number :7520001, Stockholm, Sweden
- Investigational Site Number :1580001, Taoyuan, Taiwan
- United Kingdom (2):
  - Investigational Site Number :8260001, London, London, City of
  - Investigational Site Number :8260002, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Giladi N, Alcalay RN, Cutter G, Gasser T, Gurevich T, Hoglinger GU, Marek K, Pacchetti C, Schapira AHV, Scherzer CR, Simuni T, Minini P, Sardi SP, Peterschmitt MJ. Safety and efficacy of venglustat in GBA1-associated Parkinson's disease: an international, multicentre, double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2023 Aug;22(8):661-671. doi: 10.1016/S1474-4422(23)00205-3. PMID 37479372
- [Derived] Schidlitzki A, Stanojlovic M, Fournier C, Kaufer C, Feja M, Gericke B, Garzotti M, Welford RWD, Steiner MA, Angot E, Richter F. Double-Edged Effects of Venglustat on Behavior and Pathology in Mice Overexpressing alpha-Synuclein. Mov Disord. 2023 Jun;38(6):1044-1055. doi: 10.1002/mds.29398. Epub 2023 Apr 12. PMID 37050861
- [Derived] Peterschmitt MJ, Saiki H, Hatano T, Gasser T, Isaacson SH, Gaemers SJM, Minini P, Saubadu S, Sharma J, Walbillic S, Alcalay RN, Cutter G, Hattori N, Hoglinger GU, Marek K, Schapira AHV, Scherzer CR, Simuni T, Giladi N, Sardi SP, Fischer TZ; MOVES-PD Investigators. Safety, Pharmacokinetics, and Pharmacodynamics of Oral Venglustat in Patients with Parkinson's Disease and a GBA Mutation: Results from Part 1 of the Randomized, Double-Blinded, Placebo-Controlled MOVES-PD Trial. J Parkinsons Dis. 2022;12(2):557-570. doi: 10.3233/JPD-212714. PMID 34897099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 52 sites in 16 countries. A total of 273 participants were enrolled from 15-Dec-2016 to 18-Dec-2019. Study consisted of 2 Parts: Part 1 (dose escalation period) & Part 2 (double-blind [DB] treatment period + long-term follow-up [LTFU]) period.
Pre-assignment Details: Post part 1 completion, 23 eligible & willing participants were re-randomized in Part 2 and were counted again in total enrollment number (273). i.e.,250 unique participants (29 in Part 1+221 in Part 2)+23 re-randomized in Part 2; these 23 participants are displayed only in 'participant flow' & 'adverse events' sections but not in any other section.
Groups:
- Part 1: Placebo (ROW): Participants from rest of world (ROW, except Japan), received placebo (matched to venglustat) capsule orally once daily (QD) for up to 36 weeks in Part 1.
- Part 1: Venglustat 4 mg (ROW): Participants from ROW (except Japan), received venglustat 4 milligrams (mg) capsule orally QD for up to 36 weeks in Part 1.
- Part 1: Venglustat 8 mg (ROW): Participants from ROW (except Japan), received venglustat 8 mg capsule orally QD for up to 36 weeks in Part 1.
- Part 1: Venglustat 15 mg (ROW): Participants from ROW (except Japan), received venglustat 15 mg capsule orally QD for up to 36 weeks in Part 1.
- Part 1: Placebo (Japan Only): Japanese participants received placebo (matched to venglustat) capsule orally QD for up to 52 weeks in Part 1.
- Part 1: Venglustat 4 mg (Japan Only): Japanese participants received venglustat 4 mg capsule orally QD for up to 52 weeks in Part 1.
- Part 1: Venglustat 8 mg (Japan Only): Japanese participants received venglustat 8 mg capsule orally QD for up to 52 weeks in Part 1.
- Part 1: Venglustat 15 mg (Japan Only): Japanese participants received venglustat 15 mg capsule orally QD for up to 52 weeks in Part 1.
- Part 2, DB Period: Placebo: Participants received placebo (matched to venglustat) capsule orally QD for 52 weeks in Part 2 DB period.
- Part 2, DB Period: Venglustat 15 mg: Participants received venglustat 15 mg capsule orally QD for 52 weeks in Part 2 DB period.
- Part 2, DB Period: Placebo (Re-randomized From Part 1): Participants who completed Part 1 with placebo (matched to venglustat) or venglustat 4/8/15 mg, met eligibility criteria for Part 2 and agreed to continue in the study, were re-randomized to receive placebo (matched to venglustat) capsule orally QD for 52 weeks in Part 2 DB period.
- Part 2, DB Period: Venglustat 15 mg (Re-randomized From Part 1): Participants who completed Part 1 with placebo (matched to venglustat) or venglustat 4/8/15 mg, met eligibility criteria for Part 2 and agreed to continue in the study, were re-randomized to receive venglustat 15 mg capsule orally QD for 52 weeks in Part 2 DB period.
- Part 2, LTFU Period: Placebo Then Venglustat 15 mg: Participants who were enrolled in the study in Part 2, received placebo (matched to venglustat), completed Part 2 DB period, entered long-term follow-up (LTFU) period to receive venglustat 15 mg capsule orally QD for 156 weeks.
- Part 2, LTFU Period: Venglustat 15 mg: Participants who were enrolled in the study in Part 2, received venglustat 15 mg, completed Part 2 DB period, entered LTFU period to receive venglustat 15 mg capsule orally QD for 156 weeks.
- Part 2, LTFU: Placebo Then Veng 15 mg (Re-randomized From Part 1): Participants from Part 1 who were re-randomized in the study in Part 2, received placebo (matched to venglustat) and completed Part 2 DB period, entered LTFU period to receive venglustat (Veng) 15 mg capsule orally QD for 156 weeks.
- Part 2, LTFU: Venglustat 15 mg (Re-randomized From Part 1): Participants from Part 1 who were re-randomized in the study in Part 2, received venglustat 15 mg and completed Part 2 DB period, entered LTFU period to receive venglustat 15 mg capsule orally QD for 156 weeks.
Period: Part 1: Dose Escalation Period
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only) | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg | Part 2, DB Period: Placebo (Re-randomized From Part 1) | Part 2, DB Period: Venglustat 15 mg (Re-randomized From Part 1) | Part 2, LTFU Period: Placebo Then Venglustat 15 mg | Part 2, LTFU Period: Venglustat 15 mg | Part 2, LTFU: Placebo Then Veng 15 mg (Re-randomized From Part 1) | Part 2, LTFU: Venglustat 15 mg (Re-randomized From Part 1)
Started | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 3 | 5 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Double-blind Treatment Period
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only) | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg | Part 2, DB Period: Placebo (Re-randomized From Part 1) | Part 2, DB Period: Venglustat 15 mg (Re-randomized From Part 1) | Part 2, LTFU Period: Placebo Then Venglustat 15 mg | Part 2, LTFU Period: Venglustat 15 mg | Part 2, LTFU: Placebo Then Veng 15 mg (Re-randomized From Part 1) | Part 2, LTFU: Venglustat 15 mg (Re-randomized From Part 1)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 111 | 110 | 10 | 13 | 0 | 0 | 0 | 0
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 111 | 110 | 10 | 13 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 99 | 85 | 10 | 13 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 25 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 15 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Long-term Follow-up Period
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only) | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg | Part 2, DB Period: Placebo (Re-randomized From Part 1) | Part 2, DB Period: Venglustat 15 mg (Re-randomized From Part 1) | Part 2, LTFU Period: Placebo Then Venglustat 15 mg | Part 2, LTFU Period: Venglustat 15 mg | Part 2, LTFU: Placebo Then Veng 15 mg (Re-randomized From Part 1) | Part 2, LTFU: Venglustat 15 mg (Re-randomized From Part 1)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 99 | 85 | 10 | 11 (Out of 13 completed participants in the previous part 2 DB period-arm, 2 didn't enter LTFU period.)
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 87 | 75 | 10 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 99 | 85 | 10 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 4 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Poor Compliance to Protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 64 | 7 | 8
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 8 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized unique participants (N=250) only.
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only) | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg | Total Title
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3 | 111 | 110 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (8.8) | 55.0 (3.9) | 61.0 (6.9) | 63.8 (8.7) | 52.0 (10.4) | 61.7 (5.9) | 56.7 (4.0) | 46.7 (8.1) | 59.8 (8.5) | 58.2 (9.8) | 58.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 43 | 45 | 97
  Male | 3 | 3 | 4 | 3 | 3 | 0 | 2 | 2 | 68 | 65 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 7 | 10 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 5 | 4 | 0 | 0 | 0 | 0 | 104 | 100 | 221
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and does not necessarily had to have a causal relationship with the treatment. Serious AEs (SAEs) were any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were the AEs that developed or worsened or became serious during the TEAE period (defined as the period from the time of first investigational medicinal product [IMP] administration up of 6 weeks after the last administration of the IMP).
Time Frame: From the first IMP administration up to 6 weeks after the last administration of the IMP (i.e., up to 42 weeks for ROW and up to 58 weeks for Japanese participants)
Population: Analysis was performed on safety population which included both non-Japanese (ROW) and Japanese participants who received at least 1 dose of study medication in Part 1 of the study. This outcome measure (OM) was planned to be analyzed and reported for Part 1 only and not for Part 2, as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  Any TEAE | 4 | 4 | 4 | 4 | 2 | 3 | 3 | 2
  Any TESAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 1: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included following observations/measurements: general appearance; heart, skin, respiratory auscultation; head, eyes, ears, nose, and throat, extremities/joints, and abdomen. New onset of abnormal physical examination was defined as a normal physical examination at Baseline and an abnormal physical examination during the treatment-emergent (TE) period (defined as the period from the time of first IMP administration up of 6 weeks after the last administration of the IMP). Abnormalities in physical examination were based on investigator's evaluation.
Time Frame: as for outcome 1
Population: Analysis was performed on safety population. This OM was planned to be analyzed and reported for Part 1 only and not for Part 2, as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Abnormal Neurological Examination Findings
Description: Neurological examination included at least assessments of the participant's cranial nerves, motor system (including muscle atrophy, tone, and power), mental status, deep tendon reflex, sensation, and cerebellar function. Abnormalities in neurological examination were based on investigator's evaluation.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  Abnormal cranial nerve examination | 1 | 1 | 1 | 2 | 1 | 3 | 3 | 2
  Abnormal motor examination | 3 | 4 | 4 | 3 | 3 | 3 | 3 | 3
  Abnormal strength examination | 1 | 4 | 3 | 3 | 1 | 2 | 2 | 1
  Abnormal reflex examination | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 0
  Abnormal sensory examination | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
  Abnormal coordination examination | 2 | 1 | 1 | 3 | 1 | 0 | 1 | 2
  Abnormal gait and coordination | 3 | 4 | 4 | 2 | 3 | 2 | 2 | 2

4. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Hematology
Description: Criteria for potentially clinically significant abnormalities (PCSA): Hemoglobin: less than or equal to (<=) 115 grams per liter (g/L) (Male[M]) or <=95 g/L (Female[F]), greater than or equal to (>=) 185 g/L (M) or >=165 g/L (F), Decrease from baseline (DFB) >=20 g/L; Hematocrit: <=0.37 volume/volume (v/v) (M) or <=0.32 v/v (F), >=0.55 v/v (M) or >=0.5 v/v (F); Red blood cells (RBC): >=6 Tera/L; Platelets: less than (<) 100 Giga/L, >=700 Giga/L; White blood cells (WBC): <3.0 Giga/L (Non-Black [NB]) or <2.0 Giga/L (Black [B]), >=16.0 Giga/L; Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B); Lymphocytes: <lower limit of normal (LLN), greater than (>) 4.0 Giga/L; Monocytes: <LLN, >0.7 Giga/L; Basophils: >0.1 Giga/L; Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  Hemoglobin <= 115 g/L (M); ≤ 95 g/L (F) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin >=185 g/L (M) or >=165 g/L (F) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin DFB >=20 g/L | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Hematocrit: <=0.37 v/v (M) or <=0.32 v/v (F) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Hematocrit: >=0.55 v/v (M); >=0.5 v/v (F) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC: >=6 Tera/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: <100 Giga/L | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Platelets: >=700 Giga/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC: <3.0 Giga/L (NB) or <2.0 Giga/L (B) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC: >=16.0 Giga/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils <1.5 Giga/L (NB) or <1.0 Giga/L (B) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: <LLN | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Lymphocytes: >4.0 Giga/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: <LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: >0.7 Giga/L | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Basophils: >0.1 Giga/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils >0.5 Giga/L or >ULN (ULN >=0.5 Giga/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Liver Function Parameters
Description: Criteria for PCSA: Alanine Aminotransferase (ALT): >3 ULN, >5 ULN; Aspartate aminotransferase (AST): >3 ULN; Alkaline phosphatase: >1.5 ULN; Total Bilirubin: >1.5 ULN; ALT and Bilirubin: >3 ULN and >2 ULN; Direct Bilirubin and Bilirubin: >35% and >1.5 ULN.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  ALT >3 ULN | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALT >5 ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST >3 ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST >5 ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase >1.5 ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Total Bilirubin > 1.5 ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT and Bilirubin: >3 ULN and >2 ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin and Bilirubin: >35% and >1.5 ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Renal Parameters
Description: Criteria for PCSA: Creatinine: >=150 micromoles per liter (mcmol/L) (adults), >=30% change from baseline, >=100% change from baseline; Blood urea nitrogen: >=17 millimoles (mmol)/L.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  Creatinine >=150 mcmol/L (Adults) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine >=30% change from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine >=100% change from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen >=17 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Metabolic Parameters
Description: Criteria for PCSA: Glucose: <=3.9 mmol/L and <LLN; >=11.1 mmol/L (unfasted [unfas]) or >=7 mmol/L (fasted [fas]); Albumin: <=25 g/L.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  Glucose <=3.9 mmol/L and <LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose >=11.1 mmol/L (unfas) or >=7 mmol/L (fas) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Albumin <=25 g/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Electrolytes Parameters
Description: Criteria for PCSA: Sodium: <=129 mmol/L, >=160 mmol/L; Potassium: <3 mmol/L, >=5.5 mmol/L and Chloride: <80 mmol/L, >115 mmol/L.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  Sodium <=129 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium >=160 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium <3 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium >=5.5 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride <80 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride >115 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities
Description: Criteria for PCSA: Systolic blood pressure (SBP) supine: <=95 millimeters of mercury (mmHg) and DFB >=20 mmHg; >=160 mmHg and increase from baseline (IFB) >=20 mmHg; Diastolic blood pressure (DBP) supine: <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB >=10 mmHg; SBP (Orthostatic): <=-20 mmHg; DBP (Orthostatic): <=-10 mmHg; Heart rate (HR) supine: <=50 beats per minute (bpm) and DFB >=20 bpm; >=120 bpm and IFB >=20 bpm; Weight: >=5% DFB; >=5% IFB.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  SBP (supine) <=95 mmHg and DFB >=20 mmHg | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  SBP (supine) >=160 mmHg and IFB >=20 mmHg | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  DBP (supine) <=45 mmHg and DFB >=10 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP (supine) >=110 mmHg and IFB >=10 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP (Orthostatic): <=-20 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP (Orthostatic): <=-10 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR (supine) <=50 bpm and DFB >= 20 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR (supine) >=120 bpm and IFB >=20 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight >=5% DFB | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Weight >=5% IFB | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Ophthalmological Abnormalities
Description: Clinically significant observations in left eye, right eye and any eye (any eye among left and right) were assessed by the investigator based on methods like visual acuity, slit lamp examination, examination of the cornea, lens, and retina. Any abnormal clinically significant ophthalmological examination finding (which was present at screening or not) on any eye during the treatment-emergent period corresponded to cornea verticillata, cataract and abnormal overall evaluation
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  Any eye | 3 | 3 | 4 | 2 | 2 | 3 | 3 | 0
  Right eye | 3 | 3 | 4 | 2 | 2 | 2 | 3 | 0
  Left eye | 3 | 3 | 4 | 2 | 2 | 3 | 3 | 0

11. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Electrocardiogram Abnormalities
Description: Criteria for PCSA: HR: <50 bpm; <50 bpm and DFB >=20 bpm, <40 bpm; >90 bpm, <90 bpm and IFB >=20 bpm, >100 bpm; PR Interval: >200 milliseconds (msec), >200 msec and IFB >=25%, >220 msec; QRS Interval: >110 msec, >110 msec and IFB >=25%, >120 msec; QT Interval: >500 msec; QTc Bazett (QTcB) interval: >450 msec, >480 msec, IFB >30 and <=60 msec, IFB >60 msec; QTc Fridericia (QTc F): >450 msec, >480 msec, IFB >30 and <=60 msec, IFB >60 msec.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only)
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 3 | 3 | 3 | 3
Participants
  HR: <50 bpm | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  HR: <50 bpm and DFB >=20 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR: <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR: >90 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  HR: >90 bpm and IFB >=20 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR: >100 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval: >200 msec | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  PR Interval: >200 msec and IFB >=25% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval: >220 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Interval: >110 msec | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  QRS Interval: >110 msec and IFB >=25% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Interval: >120 msec | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  QT Interval: >500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval: >450 msec | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  QTcB interval: >480 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval: IFB >30 and <=60 msec | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  QTcB interval: IFB >60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTc F: >450 msec | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  QTc F: >480 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTc F: IFB >30 and <=60 msec | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  QTc F: IFB >60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part 2: Change From Baseline to Week 52 in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II+III Total Score
Description: MDS-UPDRS is a multimodal scale consisting of 4 parts. Part II assessed motor experiences of daily living (total score range: 0 to 52). It contained 13 questions completed by the participant. Part III assessed the motor signs of PD and was administered by the rater (total score range: 0 to 132). Part III contained 33 scores based on 18 items. In both parts, higher score indicated more severe symptoms. For each question in both parts, numeric score was assigned between 0 to 4, where 0=Normal, 1=Slight, 2=Mild, 3=Moderate, 4=Severe. MDS-UPDRS Total Part II and III score = sum of Part II and III scores with score ranged from 0 (no symptom) to 184 (severe symptoms), where higher scores reflected more severe symptoms of PD. Data for this OM was not planned to be collected and analyzed for Part 1, Part 2: DB period re-randomized participants and Part 2 LTFU period, as pre-specified in protocol.
Time Frame: Baseline to Week 52
Population: Analyzed on intent-to-treat (ITT) population which included all randomized participants of Part 2 and analyzed in treatment group to which they were randomized. Here, overall number of participants analyzed = participants evaluable for this OM.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg
Number analyzed (Participants) | 95 | 81
units on a scale | 4.71 (1.27) | 7.29 (1.36)
Statistical Analysis 1: Comparison: Part 2, DB Period: Placebo vs Part 2, DB Period: Venglustat 15 mg; Least-squares (LS) mean, standard errors (SE) and p-value were estimated from mixed-effect model with repeated measures (MMRM) analysis which included fixed categorical effects of treatment group, randomization strata, time point, treatment-by-time point and strata-by-time point interaction and continuous fixed covariates Baseline value and Baseline value-by-time point interaction; Test type: Superiority; p = 0.1679, MMRM — The threshold for statistical significance was 0.05; LS mean difference = 2.58, 95% CI 2-sided [-1.10 to 6.27], Standard Error of Mean 1.87

13. Secondary Outcome: Part 2: Change From Baseline to Week 52 in Parkinson's Disease Cognitive Rating Scale (PD-CRS) Total Score
Description: The PD-CRS detects early cognitive impairment in Parkinson's disease. It is composed of 2 scales, the fronto-subcortical scale (items: sustained attention, working memory, alternating and action verbal fluency, clock drawing, immediate, and delayed free recall verbal memory) and the posterior-cortical scale (items: confrontation naming and clock copying). The total score of the fronto-subcortical scale (sum of all items) ranged from 0 (worst) to 104 (maximum score indicates better) and the total score of the posterior-cortical scale (sum of all items) ranged from 0 (worst) to 30 (maximum score indicates better). The PD-CRS Total score = the sum of PD-CRS fronto-subcortical score and the PD-CRS posterior-cortical score, which ranged from 0 to 134, where higher score = less impairment.
Time Frame: Baseline to Week 52
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed = participants evaluable for this OM. Data for this OM was not planned to be collected and analyzed for Part 1, Part 2: DB period re-randomized participants and Part 2 LTFU period, as pre-specified in protocol.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg
Number analyzed (Participants) | 94 | 82
units on a scale | 0.32 (1.27) | -0.65 (1.35)
Statistical Analysis 1: Comparison: Part 2, DB Period: Placebo vs Part 2, DB Period: Venglustat 15 mg; LS mean, SE and P-value were estimated from MMRM analysis which included fixed categorical effects of treatment group, randomization strata, time point, treatment-by-time point and strata-by-time point interaction and continuous fixed covariates Baseline value and Baseline value-by-time point interaction; Test type: Superiority; p = 0.5996, MMRM — The threshold for statistical significance was 0.05; LS mean difference = -0.97, 95% CI 2-sided [-4.63 to 2.68], Standard Error of Mean 1.85

14. Secondary Outcome: Part 2: Change From Baseline to Week 52 in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I+ II+III Score
Description: MDS-UPDRS is a multimodal scale consisting of 4 parts. Part I assessed non-motor experiences of daily living and has 2 components (total score range: 0 to 52): Part IA contained 6 questions and was assessed by the examiner (total score range: 0 to 24). Part IB contained 7 questions on non-motor experiences of daily living which was completed by the participant (total score range: 0 to 28). Part II (13 questions completed by the participant) assessed motor experiences of daily living (total score range: 0 to 52). Part III assessed motor signs of PD and was administered by the rater (total score range: 0 to 132). Part III contained 33 scores based on 18 items. In all parts, higher score indicated more symptoms. For each question, numeric score was assigned between 0 to 4, where 0=Normal, 1=Slight, 2=Mild, 3=Moderate, 4=Severe. MDS-UPDRS total score = sum of Parts I, II, and III (Range: 0 to 236). Higher score = more severe symptoms of PD.
Time Frame: Baseline to Week 52
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg
Number analyzed (Participants) | 95 | 81
units on a scale | 5.87 (1.45) | 9.99 (1.55)
Statistical Analysis 1: Comparison: Part 2, DB Period: Placebo vs Part 2, DB Period: Venglustat 15 mg; LS mean, SE and P-value were estimated from MMRM analysis which included fixed categorical effects of treatment group, randomization strata, time point, treatment-by-time point and strata-by-time point interaction and continuous fixed covariates Baseline value and Baseline value-by-time-interaction; Test type: Superiority; p = 0.0535, MMRM — The threshold for statistical significance was 0.05; LS mean difference = 4.13, 95% CI 2-sided [-0.06 to 8.32], Standard Error of Mean 2.13

15. Secondary Outcome: Part 2: Change From Baseline to Week 52 in Hoehn and Yahr (H and Y) Score
Description: H and Y scale measured how Parkinson's symptoms progress and the level of disability. Scale allocated stage scores were from 0 to 5 to indicate relative level of disability as: Stage 0: no symptoms; Stage 1: symptoms on one side of the body only; Stage 2: symptoms on both sides of the body, without impairment of balance; Stage 3: Mild to moderate bilateral disease; some postural instability; physically independent; Stage 4: Severe disability; still able to walk or stand unassisted and Stage 5: Wheelchair bound or bedridden unless aided, where higher stage score described an increased severity of disease.
Time Frame: Baseline to Week 52
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg
Number analyzed (Participants) | 95 | 80
units on a scale | 0.18 (0.05) | 0.20 (0.06)
Statistical Analysis 1: Comparison: Part 2, DB Period: Placebo vs Part 2, DB Period: Venglustat 15 mg; LS mean, SE and P-value: estimated from MMRM analysis which included fixed categorical effects of treatment group, randomization strata, time point, treatment-by-time point and strata-by-time point interaction and continuous fixed covariates Baseline value and Baseline value-by-time-interaction; Test type: Superiority; p = 0.7400, MMRM — The threshold for statistical significance was 0.05; LS mean difference = 0.03, 95% CI 2-sided [-0.12 to 0.17], Standard Error of Mean 0.08

ADVERSE EVENTS:
Time Frame: From the first IMP administration up to 6 weeks after the last administration of the IMP (i.e., in Part 1: up to 42 weeks for ROW, up to 58 weeks for Japanese participants; in Part 2 DB period: up to 60 weeks; in Part 2 LTFU period: up to 164 weeks).
Description: Reported AEs and deaths were TEAEs that developed/worsened in grade or became serious during TEAE period (defined as the time from the first dose of the IMP to the last dose of IMP + 6 weeks). Analysis was performed on safety population.
Arm/Group | Part 1: Placebo (ROW) | Part 1: Venglustat 4 mg (ROW) | Part 1: Venglustat 8 mg (ROW) | Part 1: Venglustat 15 mg (ROW) | Part 1: Placebo (Japan Only) | Part 1: Venglustat 4 mg (Japan Only) | Part 1: Venglustat 8 mg (Japan Only) | Part 1: Venglustat 15 mg (Japan Only) | Part 2, DB Period: Placebo | Part 2, DB Period: Venglustat 15 mg | Part 2, DB Period: Placebo (Re-randomized From Part 1) | Part 2, DB Period: Venglustat 15 mg (Re-randomized From Part 1) | Part 2, LTFU Period: Placebo Then Venglustat 15 mg | Part 2, LTFU Period: Venglustat 15 mg | Part 2, LTFU: Placebo Then Veng 15 mg (Re-randomized From Part 1) | Part 2, LTFU: Venglustat 15 mg (Re-randomized From Part 1)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/4 | 0/3 | 0/3 | 0/3 | 0/3 | 0/111 | 1/110 | 0/10 | 0/13 | 1/87 | 0/75 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/4 | 0/3 | 0/3 | 0/3 | 0/3 | 12/111 | 12/110 | 0/10 | 3/13 | 15/87 | 9/75 | 3/10 | 1/11
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/5 | 4/4 | 2/3 | 3/3 | 3/3 | 2/3 | 87/111 | 95/110 | 8/10 | 11/13 | 53/87 | 39/75 | 7/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (ROW) (N=4) | Part 1: Venglustat 4 mg (ROW) (N=4) | Part 1: Venglustat 8 mg (ROW) (N=5) | Part 1: Venglustat 15 mg (ROW) (N=4) | Part 1: Placebo (Japan Only) (N=3) | Part 1: Venglustat 4 mg (Japan Only) (N=3) | Part 1: Venglustat 8 mg (Japan Only) (N=3) | Part 1: Venglustat 15 mg (Japan Only) (N=3) | Part 2, DB Period: Placebo (N=111) | Part 2, DB Period: Venglustat 15 mg (N=110) | Part 2, DB Period: Placebo (Re-randomized From Part 1) (N=10) | Part 2, DB Period: Venglustat 15 mg (Re-randomized From Part 1) (N=13) | Part 2, LTFU Period: Placebo Then Venglustat 15 mg (N=87) | Part 2, LTFU Period: Venglustat 15 mg (N=75) | Part 2, LTFU: Placebo Then Veng 15 mg (Re-randomized From Part 1) (N=10) | Part 2, LTFU: Venglustat 15 mg (Re-randomized From Part 1) (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subacute Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anastomotic Leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative Delirium (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Freezing Phenomenon (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
On And Off Phenomenon (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0)
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive Urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (ROW) (N=4) | Part 1: Venglustat 4 mg (ROW) (N=4) | Part 1: Venglustat 8 mg (ROW) (N=5) | Part 1: Venglustat 15 mg (ROW) (N=4) | Part 1: Placebo (Japan Only) (N=3) | Part 1: Venglustat 4 mg (Japan Only) (N=3) | Part 1: Venglustat 8 mg (Japan Only) (N=3) | Part 1: Venglustat 15 mg (Japan Only) (N=3) | Part 2, DB Period: Placebo (N=111) | Part 2, DB Period: Venglustat 15 mg (N=110) | Part 2, DB Period: Placebo (Re-randomized From Part 1) (N=10) | Part 2, DB Period: Venglustat 15 mg (Re-randomized From Part 1) (N=13) | Part 2, LTFU Period: Placebo Then Venglustat 15 mg (N=87) | Part 2, LTFU Period: Venglustat 15 mg (N=75) | Part 2, LTFU: Placebo Then Veng 15 mg (Re-randomized From Part 1) (N=10) | Part 2, LTFU: Venglustat 15 mg (Re-randomized From Part 1) (N=11)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Borderline Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract Cortical (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 4 (5) | 1 (1) | 1 (2) | 5 (6) | 3 (4) | 0 (0) | 0 (0)
Cataract Nuclear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 9 (9) | 1 (1) | 1 (1) | 11 (11) | 4 (4) | 0 (0) | 2 (2)
Corneal Infiltrates (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema Eyelids (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 23 (25) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 1 (1) | 0 (0)
Cyclic Vomiting Syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 8 (9) | 23 (27) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 9 (12) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 12 (13) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 11 (11) | 10 (13) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulpitis Dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Retinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea Pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 11 (17) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (24) | 10 (12) | 0 (0) | 1 (4) | 9 (12) | 2 (3) | 0 (0) | 3 (3)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Procedural Nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 9 (14) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Extremity Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorea (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 12 (14) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 15 (20) | 22 (31) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hyperreflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 8 (8) | 0 (0) | 2 (2) | 11 (11) | 4 (4) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radial Nerve Palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Resting Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless Legs Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep Deficit (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 8 (9) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 5 (5) | 0 (0) | 2 (2) | 7 (7) | 2 (3) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 9 (10) | 1 (1) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Drug Abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hallucination, Visual (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Impulsive Behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 6 (6) | 9 (10) | 0 (0) | 0 (0) | 5 (6) | 3 (3) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poor Quality Sleep (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rapid Eye Movement Sleep Behaviour Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertonic Bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ovarian Failure (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 10 (11) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar Cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study did not achieve its primary or secondary endpoints at the time of the analysis of the double-blind 52-week treatment period of Part 2 and was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT02906020/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02906020/SAP_001.pdf